CLINICAL TRIAL: NCT05091983
Title: Restrictive Eating Disorders: From Childhood Orality Disorder to Adolescent Dysensoriality (Orality Dysensoriality and Eating Disorder)
Brief Title: Restrictive Eating Disorders: From Childhood Orality Disorder to Adolescent Dysensoriality
Acronym: ODYSSED
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211140; 2021-A01755-36 (Other: France : ANSM)
Record Dates: First submitted 2021-09-27; First posted 2021-10-25 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Eating Disorders in Adolescence; Avoidant Restrictive Food Intake Disorder
Keywords: Restrictive eating disorder; anorexia nervosa; Avoidant/Restrictive Food Intake Disorder; sensory modulation disorder; sensory modulation symptoms; sensory over responsivity; sensory integration
MeSH Terms: conditions — Avoidant Restrictive Food Intake Disorder; Anorexia Nervosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Restrictive eating disorder group: Adolescents between 12 and 18 y.o. Restrictive eating disorders diagnosis (Anorexia Nervosa or ARFID) answering DSM-5 criteria
  Interventions: Other: Sensory Processing Scale Inventory (SPSI); Other: Autism Spectrum Screening Quotient (ASSQ); Other: GAD 7; Other: Conners abridged; Other: EAT 26
- Control group: Adolescents between 12 and 18 y.o. No eating disorders
  Interventions: Other: Sensory Processing Scale Inventory (SPSI); Other: Autism Spectrum Screening Quotient (ASSQ); Other: GAD 7; Other: Conners abridged

INTERVENTIONS:
Other: Sensory Processing Scale Inventory (SPSI) — The Sensory Processing Scale Inventory (SPSI) is the main questionnaire. It allows to define over and under sensitive profiles. It's a self-administrated questionnaire
Other: Autism Spectrum Screening Quotient (ASSQ) — The ASSQ allows to detect autism spectrum disorders (ASD). This quotient is proposed to the group because the investigators know that ASD are often correlated with sensory integration disorders.
  It's answered by the participant's parents.
Other: GAD 7 — The GAD7 questionnaire allows to detect anxiety disorder. This questionnaire is proposed to the group because the investigators know that anxiety disorders are often correlated with sensory integration disorders.
  It's a self-administrated questionnaire.
Other: Conners abridged — The Conners abridged questionnaire allows to detect attention-deficit hyperactivity disorder (ADHD). This questionnaire is proposed to the group because the investigators know that ADHD are often correlated with sensory integration disorders.
  The questionnaire is answered by the participant's parents.
Other: EAT 26 — The EAT 26 questionnaire allows to detect anorexia nervosa. It is proposed to the patient with an eating disorder to establish the level of severity of their disease.
  It's a self-administrated questionnaire.
  Groups: Restrictive eating disorder group

SUMMARY:
This study offers to determine whether adolescent patients with a restrictive eating disorder have variations in their sensoriality compared to a control group.

DETAILED DESCRIPTION:
Eating disorders are a frequent reason for consultation in pediatrics at all ages.

When they are small, children may have an orality disorder. There are multiple potential causes for this disorder: psychogenic, oropraxic but also sensory. The treatment is then adapted to the patient, with, among other things, an orientation towards professionals trained in sensory disorders.

As they grow up, adolescents are particularly at risk of developing eating disorders, which are pathologies that correspond to a biopsychosocial model of understanding that includes psychogenetic, neuroendocrine and immune factors.

Despite major advances in the understanding of this disease, the sensory dimension for these patients is still little studied and is not taken into account in the treatment proposed to adolescents suffering from eating disorders.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent between 12 to 18 years old.
* Non-opposition of the adolescent and his or her legal guardians collected before the start of the study.
* Patient group: Diagnosis of restrictive eating disorders (Anorexia Nervosa typical or atypical, ARFID) meeting DSM-5 criteria.
* Control group: absence of eating disorders.

Exclusion Criteria:

* Eating disorders secondary to another psychiatric pathology.
* Precarious health status with somatic and/or psychiatric instability that does not allow to answer the questionnaire.
* Language barrier.
* Opposition of the adolescent and/or his/her legal representatives obtained before the start of the study
* Patient under " AME " (medical state help)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The participants were all recruited at the Maison de Solenn, Cochin - Paris, a service specialized in the treatment of eating disorders for adolescents. The participants in the control group are patients followed in this center for another reason than an eating disorder. The participants were recruited in consultation, in day hospital or in complete hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Average Sensory Processing Scale Inventory (SPSI) scores between the two groups | Inclusion
  Comparison of average Sensory Processing Scale Inventory (SPSI) scores between the two groups This questionnaire focuses on sensoriality. It allows the definition of over or under-reactive sensory profiles. It is made of two lists (list #1 : 73 items ; list #2 : 29 items).
  The SPSI questionnaire is in English. For this reason, a group of experts from La Maison de Solenn met to translate it into French being as faithful as possible to the original questionnaire. Each checklist has its own score, the result is the sum of the points obtained (one point for YES, zero points for NO) (6).
  Two groups will be formed: a group with eating disorders and a control group. The questionnaire will be answered only once and will be proposed to the participant at the end of a consultation at the Maison de Solenn for his usual follow-up or during a hospitalization (full time hospitalization or in day hospital).

SECONDARY OUTCOMES:
Screening for pathologies known to be associated with a sensory disorder | Inclusion
  Screening questionnaires for Autism Spectrum Disorder (ASD) will be distributed in order to identify disorders associated with a particular sensory profile. This will allow statistical results to be refined by performing multivariate analyses.
Screening for pathologies known to be associated with a sensory disorder | Inclusion
  Screening questionnaires for Attention Deficit Hyperactivity Disorder (ADHD) will be distributed in order to identify disorders associated with a particular sensory profile. This will allow statistical results to be refined by performing multivariate analyses.
Screening for pathologies known to be associated with a sensory disorder | Inclusion
  Screening questionnaires for Generalized Anxiety Disorder (GAD) will be distributed in order to identify disorders associated with a particular sensory profile. This will allow statistical results to be refined by performing multivariate analyses.
Search for a link between the eating disorders severity and sensory disorders | Inclusion
  The EAT 26 questionnaire is used to measure the severity of an eating disorder. It will be proposed only to the participants of the eating disorder group.
  This measure of severity will assess whether there is a relationship between the severity of the ED and the severity of the sensory disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Corinne BLANCHET, Principal Investigator — APHP - Cochin Hospital
Locations (1):
- Maison de Solenn Maison des Adolescents, Cochin Hospital, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Battle DE. Diagnostic and Statistical Manual of Mental Disorders (DSM). Codas. 2013;25(2):191-2. doi: 10.1590/s2317-17822013000200017. No abstract available. PMID 24413388
- [Background] Gorwood P, Blanchet-Collet C, Chartrel N, Duclos J, Dechelotte P, Hanachi M, Fetissov S, Godart N, Melchior JC, Ramoz N, Rovere-Jovene C, Tolle V, Viltart O, Epelbaum J. New Insights in Anorexia Nervosa. Front Neurosci. 2016 Jun 29;10:256. doi: 10.3389/fnins.2016.00256. eCollection 2016. PMID 27445651
- [Background] Schoen SA, Miller LJ, Green KE. Pilot study of the Sensory Over-Responsivity Scales: assessment and inventory. Am J Occup Ther. 2008 Jul-Aug;62(4):393-406. doi: 10.5014/ajot.62.4.393. PMID 18712002
- See also: LEBLANC V, LECOUFLE A, BOURGEOIS C, al et. Boîte à idées pour oralité malmenée du jeune enfant [Internet]. Nutricia; s. d. 19 p — https://www.google.fr/url?sa=t&rct=j&q=&esrc=s&source=web&cd=1&cad=rja&uact=8&ved=0ahUKEwi7kMTQhq7UAhUGXhQKHY36ACQQFggnMAA&url=http%3A%2F%2Fpontt.net%2Fwp-content%2Fuploads%2F2014%2F02%2Fboite-a-idee_oralite.pdf&usg=AFQjCNEtleesHBaMo8fal--N4WA1W7VVLQ&sig2=WmsCcW61RyWvGV8szKxwyg